CLINICAL TRIAL: NCT06061536
Title: A Randomized, Controlled, Open-label, Dose-exploration Study to Assess the Effectiveness and Safety of Lipovirtide Combined With Nucleoside Drugs in HIV-infected Patients Who Have Not Received Antiviral Treatment Before.
Brief Title: Assess the Effectiveness and Safety of Lipovirtide Combined With Nucleoside Drugs in HIV-infected Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanxi Kangbao Biological Product Co., Ltd. (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SXKB-LP-80-201
Record Dates: First submitted 2023-09-18; First posted 2023-09-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: HIV
Keywords: Lipovirtide; HIV; nucleoside drugs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A：Lipovirtide 10mg+3TC+TDF (Experimental): Lipovirtide 10mg+3TC+TDF（LP-80：once a week；3TC+TDF：once daily）
  Interventions: Drug: Lipovirtide 10mg
- Group B：Lipovirtide 40mg+3TC+TDF (Experimental): Lipovirtide 40mg+3TC+TDF（LP-80：once a week；3TC+TDF：once daily）
  Interventions: Drug: Lipovirtide 40mg
- Group C：Lipovirtide 60mg+3TC+TDF (Experimental): Lipovirtide 60mg+3TC+TDF（LP-80：once every 2 weeks；3TC+TDF：once daily）
  Interventions: Drug: Lipovirtide 60mg
- Group D：DTG +3TC + TDF (Experimental): DTG +3TC + TDF（once daily）
  Interventions: Drug: DTG

INTERVENTIONS:
Drug: Lipovirtide 10mg — Lipovirtide 10mg+3TC+TDF（LP-80：once a week；3TC+TDF：once daily）；
  Other Names: 3TC; TDF
  Arms: Group A：Lipovirtide 10mg+3TC+TDF
Drug: Lipovirtide 40mg — Lipovirtide 40mg+3TC+TDF（LP-80：once a week；3TC+TDF：once daily）；
  Other Names: 3TC; TDF
  Arms: Group B：Lipovirtide 40mg+3TC+TDF
Drug: Lipovirtide 60mg — Lipovirtide 60mg+3TC+TDF（LP-80：once every 2 weeks；3TC+TDF：once daily）；
  Other Names: 3TC; TDF
  Arms: Group C：Lipovirtide 60mg+3TC+TDF
Drug: DTG — DTG +3TC + TDF（once daily）.
  Other Names: 3TC; TDF
  Arms: Group D：DTG +3TC + TDF

SUMMARY:
A randomized, controlled, open-label, dose-exploration study to assess the effectiveness and safety of Lipovirtide combined with nucleoside drugs in HIV-infected patients who have not received antiviral treatment before.

DETAILED DESCRIPTION:
multiple sites, randomized, open-label, controlled study design. 64 eligible subjects will be enrolled in this study, and they will be randomly assigned to each group in a 1:1:1:1 proportion, 16 subjects in each group. Each site will compete to enroll subjects.

The 4 groups are as follows： Group A：Lipovirtide 10mg+3TC+TDF（LP-80：once a week；3TC+TDF：once daily）； Group B：Lipovirtide 40mg+3TC+TDF（LP-80：once a week；3TC+TDF：once daily）； Group C：Lipovirtide 60mg+3TC+TDF（LP-80：once every 2 weeks；3TC+TDF：once daily）； Group D：DTG +3TC + TDF（once daily）.

ELIGIBILITY:
Inclusion Criteria:

1. age≥18 years (including the critical value) when signed the informed consent form ,.male or female.
2. Untreated, confirmed HIV-1 infected patients;
3. HIV RNA viral load≥1000 copies/mL；
4. CD4+ T cell counts≥200 cells/mm3；
5. Subjects who have no plans for conception within the 2 weeks prior to screening and 3 months after the end of the trial, and who agree to use effective non-pharmacological contraceptive measures during the trial;
6. Sign informed consent prior to the test and fully understand the purpose, nature, methods, and possible adverse reactions, and be willing to participate in the study.

Exclusion Criteria:

1. Subjects with an allergy history or hypersensitivity to any component or excipient of the investigational drug;
2. Subjects with severe opportunistic infections or opportunistic tumors;
3. Subjects with confirmed AIDS or in the acute infection stage;
4. Hepatitis B virus surface antigen (HBsAg)/hepatitis C virus antibody (HCV-Ab) Positive;
5. ALT and/or AST≥5×ULN；
6. ALT≥3×ULN and total bilirubin≥2×ULN (direct bilirubin/total bilirubin>35%;
7. GFR<70ml/min/1.73m2 (estimated from creatinine values based on the CKD-EPI Creatinine 2009 Equation), or creatinine ≥ULN;
8. Subjects with severe and uncontrolled chronic diseases, metabolic diseases, neurological and psychiatric diseases;
9. Subjects with a pancreatitis disease history ever before;
10. Subjects who are pregnant or lactating women;
11. Subjects with a history of drug abuse, alcoholism, or substance misuse;
12. Any clinical trials in the 3 months prior to the screening of the trial; 13）Subjects may not be able to complete this study or other investigators' judgment for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
HIV-1 RNA <50 copies/ml | at Day 169 after receiving Lipovirtide administration.
  The proportion of subjects with HIV-1 RNA <50 copies/ml at Day 169 after receiving Lipovirtide administration.

SECONDARY OUTCOMES:
HIV-1 RNA <50 copies/ml | at Day 29、Day 85、Day 169 after receiving Lipovirtide administration
  The proportion of subjects with HIV-1 RNA <50 copies/ml at Day 29、Day 85、Day 169 after receiving Lipovirtide administration
HIV-1 RNA <400 copies/ml | at Day 85、Day 169 after receiving Lipovirtide administration
  The proportion of subjects with HIV-1 RNA <400 copies/ml at Day 85、Day 169 after receiving Lipovirtide administration
CD4+ T-cell and CD8+ T-cell | at Day 85 and Day 169 after receiving Lipovirtide administration
  The changes in CD4+ T-cell and CD8+ T-cell counts compared to baseline at Day 85 and Day 169 after receiving Lipovirtide administration
HIV-1 RNA <50 copies/ml | Within Day 169 of after receiving Lipovirtide administration
  The time required to achieve viral suppression (HIV-1 RNA <50 copies/ml)
HIV-1 RNA | Within Day 169 of after receiving Lipovirtide administration
  The temporal changes in log-transformed HIV-1 RNA levels compared to baseline
Changes from baseline in respiration rate of Vital Signs | Within Day 169 of after receiving Lipovirtide administration
  Respiration rate in times / minute
Changes from baseline in blood pressure of Vital Signs | Within Day 169 of after receiving Lipovirtide administration
  Blood pressure in mmHg
Changes from baseline in body temperature of Vital Signs | Within Day 169 of after receiving Lipovirtide administration
  Body temperature in Celsius degree
Changes from baseline in ECG PR intervalThe cardiac rhythm is showed in 12 Leads | Within Day 169 of after receiving Lipovirtide administration
  Ambulatory Electrocardiogram in the form of continuous curve. Changes of this continuous curve will be recorded.
Changes from baseline in ECG QRS intervalThe cardiac rhythm is showed in 12 Leads | Within Day 169 of after receiving Lipovirtide administration
  Ambulatory Electrocardiogram in the form of continuous curve. Changes of this continuous curve will be recorded
Changes from baseline in ECG QT intervalThe cardiac rhythm is showed in 12 Leads | Within Day 169 of after receiving Lipovirtide administration
  Ambulatory Electrocardiogram in the form of continuous curve. Changes of this continuous curve will be recorded
Changes from baseline in Blood lactate of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of blood lactate will be recorded
Changes from baseline in Pregnancy test of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Pregnancy test will be tested in female subjects
Changes from baseline in red blood cell count of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Red blood cell count in whole blood is reported in the form of number
Changes from baseline in white blood cell count of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  White blood cell count in whole blood is reported in the form of number
Changes from baseline in neutrophil count of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Neutrophil count in whole blood is reported in the form of number
Changes from baseline in lymphocyte count of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Lymphocyte count in whole blood is reported in the form of number
Changes from baseline in platelet count of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Platelet count in whole blood is reported in the form of number.
Changes from baseline in hemoglobin of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of hemoglobin concentration（g/dL）in whole blood will be recorded.
Changes from baseline in PT of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Prothrombin time (PT) is a screening test for exogenous coagulation factors
Changes from baseline in INR of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  International standardized ratio (INR) is calculated from prothrombin time and international sensitivity index (ISI) of the reagent
Changes from baseline in APTT of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of total bilirubin concentration (μmol/L) in serum will be recorded
Changes from baseline in direct bilirubin of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of direct bilirubin concentration (μmol/L) in serum will be recorded.
Changes from baseline in ALT of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of ALT concentration (U/L) in serum will be recorded
Changes from baseline in AST of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of AST concentration (U/L) in serum will be recorded
Changes from baseline in total protein of Laboratory Examination. | Within Day 169 of after receiving Lipovirtide administration
  Changes of total protein concentration (g/L) in serum will be recorded.
Changes from baseline in albumin of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of albumin concentration (g/L) in serum will be recorded
Changes from baseline in creatinine of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of creatinine concentration (μmol/L) in serum will be recorded
Changes from baseline in glucose of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of glucose concentration (mmol/L) in serum will be recorded.
Changes from baseline in potassium of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of potassium concentration (mmol/L) in serum will be recorded
Changes from baseline in sodium of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of sodium concentration (mmol/L) in serum will be recorded
Changes from baseline in chlorine of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of chlorine concentration (mmol/L) in serum will be recorded
Changes from baseline in urine specific gravity of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of urine specific gravity will be recorded.
Changes from baseline in urine pH of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of urine pH value will be recorded
Changes from baseline in urine glucose of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of urine glucose will be examined by qualitative test (positive or negative
Changes from baseline in urine protein of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of urine protein will be examined by qualitative test (positive or negative
Changes from baseline in urine ketone body of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of urine ketone body will be examined by qualitative test (positive or negative).
Changes from baseline in urine white blood cell of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of white blood cell in urine will be examined by qualitative test (positive or negative).
Changes from baseline in urine occult blood of Laboratory Examination. | Within Day 169 of after receiving Lipovirtide administration
  Changes of urine occult blood will be examined by qualitative test (positive or negative)
Changes from baseline in LDH of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of LDH concentration (U/L) in serum will be recorded.
Changes from baseline in Triglyceride of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of Triglyceride concentration (mmol/L) in serum will be recorded
Changes from baseline in ALP of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of ALP concentration (U/L) in serum will be recorded
Changes from baseline in CHOL of Laboratory Examination | Within Day 169 of after receiving Lipovirtide administration
  Changes of CHOL concentration (mmol/L) in serum will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Ping Ma, Doctor, Study Director — Tianjin Second People's Hospital
Locations (1):
- Tianjin Second People's Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No